CLINICAL TRIAL: NCT03507062
Title: Effect of Crystalloids With Different SID on Hemodilution, Plasmatic Acid Base Equilibrium and Urinary Electrolytes in Patients During General Anesthesia
Brief Title: Effect of Crystalloids With Different SID on pH, and Urinary Electrolytes During General Anesthesia
Acronym: CRYSID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Cristina Dominedò (Unknown); Marco Rossi (Unknown); Rossano Festa (Unknown); Nicoletta Filetici (Unknown); Marta Cicetti (Unknown); Domenico Luca Grieco (Unknown); Massimo Antonelli (Unknown)
Responsible Party: Principal Investigator, Antonio Maria Dell'Anna, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1669
Record Dates: First submitted 2018-03-15; First posted 2018-04-24 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: SID; Acid-Base Imbalance
Keywords: pH; crystalloids
MeSH Terms: conditions — Sudden Infant Death; Acid-Base Imbalance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chloride-rich solution (Experimental): Patients will receive two boluses of 10 and 20 ml/kg of the 0.9% saline in two different moments after at least 1 hour from each other. Plasma arterial blood gas (ABG) and electrolytes, along with plasmatic creatinine, albumin and phosphate will be measured immediately before and five minutes after fluid boluses. Urinary electrolytes (Na, K, Cl) will be measured immediately before fluid bolus and after one hour from fluid administration along with ABG and plasmatic electrolytes and creatinine, phosphate and albumin.
  Interventions: Other: 0.9% saline administration
- Low-chloride solution A (Experimental): Patients will receive two boluses of 10 and 20 ml/kg of Ringer's lactate in two different moments after at least 1 hour from each other. Plasma arterial blood gas (ABG) and electrolytes, along with plasmatic creatinine, albumin and phosphate will be measured immediately before and five minutes after fluid boluses. Urinary electrolytes (Na, K, Cl) will be measured immediately before fluid bolus and after one hour from fluid administration along with ABG and plasmatic electrolytes and creatinine, phosphate and albumin.
  Interventions: Other: Ringer's lactate administration
- Very low-chloride solution (Experimental): Patients will receive two boluses of 10 and 20 ml/kg of a plasmalyte-like solution (namely soluzione elettrolitica reintegrante [SER]) in two different moments after at least 1 hour from each other. Plasma arterial blood gas (ABG) and electrolytes, along with plasmatic creatinine, albumin and phosphate will be measured immediately before and five minutes after fluid boluses. Urinary electrolytes (Na, K, Cl) will be measured immediately before fluid bolus and after one hour from fluid administration along with ABG and plasmatic electrolytes and creatinine, phosphate and albumin.
  Interventions: Other: Plasmalyte-like solution administration

INTERVENTIONS:
Other: 0.9% saline administration — Each patient will receive 0.9%saline based on attending physician decision
  Arms: Chloride-rich solution
Other: Ringer's lactate administration — Each patient will receive Ringer's lactate based on attending physician decision
  Arms: Low-chloride solution A
Other: Plasmalyte-like solution administration — Each patient will receive Plasmalyte-like solution based on attending physician decision
  Arms: Very low-chloride solution

SUMMARY:
The present study will investigate variations in acid base equilibrium caused by the administration of four different crystalloids with increasing strong ion difference (0.9% saline, Ringer's lactate, Ringer's acetate, plasmalyte-like solution) in patients during general anesthesia.

The same crystalloid will be administered throughout the surgery. In order to assess the effect of hemodilution, every patient will receive two fluid boli with different volumes of the same solution. pH and strong ion variations, togher with the renal response to acid base disturbances, will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (between 18 and 75 years old);
* ASA (American Society of Anesthesiologists) physical status classification system 1 or 2;
* Patients undergoing spinal surgery under general anesthesia, intubated and mechanically ventilated;
* Normal preoperative albumin;
* Surgery with an estimated duration of at least 3 hours.

Exclusion Criteria:

* Patients who are pregnant;
* Patients with obesity (BMI > 35);
* Patients with a chronic obstructive pulmonary disease (COPD);
* Patients with obstructive sleep apnea (OSA) treated with CPAP;
* Patients with chronic heart failure (CHF) with a NYHA (New York Heart Association) class ≥2;
* Patients receiving diuretics in the pre-operative period;
* Patients with a chronic kidney disease (CKD), defined as a GFR < 60 ml/min/1.73 m2;
* Patients with diabetes mellitus treated with insulin;
* Patients with myopathies; Patients undergoing a surgery with likely fluid losses or with unexpected bleeding during surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
pH modification | Surgery
  The primary outcome of this physiological study is to evaluate, in vivo, the effect of crystalloid administration with different SID on acid base equilibrium, in particular pH variations will be considered.

SECONDARY OUTCOMES:
Urinary SID modification (mEq/L) after crystalloids administration with different SID and chloride load | Surgery
  renal response to acid base disturbances caused by different crystalloid infusions and different volumes.
SID and plasmatic weak acid (A tot) variations measured in mEq/L | Surgery
  We will explore the changes in apparent SID (SIDapp) and effective SID (SIDeff) and strong ion gap (SIG), as well as A tot after administration of solutions with different SID

CONTACTS AND LOCATIONS:
Overall Officials: Antonio M Dell'Anna, MD, Principal Investigator — Fondazione Policlinico A. Gemelli
Locations (1):
- Fondazione Policlinico A. Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dell'Anna AM, Grieco DL, Dominedo C, Cicetti M, Cisterna I, Festa R, Lamacchia R, Gianni G, Filetici N, Michi T, Rossi C, Alcaro FD, Mele A, Rocchi A, Del Prete D, Meluzio MC, Tamburrelli FC, Rossi M, Antonelli M. Stewart's theory and acid-base changes induced by crystalloid infusion in humans: a randomized physiological trial. Ann Intensive Care. 2025 Apr 22;15(1):54. doi: 10.1186/s13613-025-01473-9. PMID 40263186